CLINICAL TRIAL: NCT00766285
Title: Safety and Immunogenicity of High Dose Baculovirus-Expressed Recombinant Trivalent HA Influenza Vaccine in Adult Recipients of Allogeneic Hematopoietic Stem Cell Transplantation: Phase II Double-Blind Trial
Brief Title: High Dose Influenza in Immunosuppressed Subjects
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 06-0069
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2009-12

CONDITIONS: Influenza
Keywords: Baculovirus, influenza, stem cell transplant
MeSH Terms: conditions — Influenza, Human | interventions — trivalent baculovirus-expressed influenza-virus hemagglutinin vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- TIV (Active Comparator): 50 subjects to receive 45 mcg of TIV administered on Day 0 and Day 28.
  Interventions: Biological: Trivalent inactivated influenza vaccine
- rHAO (Experimental): 50 subjects to receive 405 mcg of rHAO administered on Day 0 and Day 28.
  Interventions: Biological: Trivalent Baculovirus-expressed Influenza HA vaccine

INTERVENTIONS:
Biological: Trivalent inactivated influenza vaccine — Standard trivalent influenza vaccine consisting of 15 mcg per antigen (45 mcg total) by intramuscular deltoid injection.
  Arms: TIV
Biological: Trivalent Baculovirus-expressed Influenza HA vaccine — Influenza virus hemagglutinin proteins expressed in insect (SF+) cells under serum free conditions by recombinant baculovirus.
  Arms: rHAO

SUMMARY:
Influenza is a common infection of the upper airways and lungs, and is caused by viruses. Cancer patients may need a stronger influenza vaccine than the general population to protect against influenza. The experimental vaccine is designed to be 9 times stronger than the standard vaccine, which may cause a stronger immune response against influenza in patients with a weakened immune system. The goal of this study is to compare the effects of a new experimental influenza vaccine to the effects of the standard influenza vaccine. One hundred bone marrow recipients, adult volunteers from the MD Anderson Cancer Center, 18 years of age or older, will participate in this study. They will be randomly (by chance) assigned to receive 2 doses of either the standard licensed influenza vaccine or the experimental influenza vaccine. Participants will be asked to complete 5 study visits and 3 telephone contacts. Study procedures include blood draws. The duration of participation is about 6 months.

DETAILED DESCRIPTION:
Bone marrow transplantation (BMT) patients are immunocompromised to a varying degree depending upon genetic relationship between donor and recipient with compromising therapy required for allogeneic transplants. Responses to influenza vaccine in this population have been poor and yet influenza virus infection can lead to serious disease. There is a need for prophylaxis against influenza in this population. One approach to improving immune responses to influenza vaccines in BMT patients could be to increase dosage and number of doses of vaccine. This approach has increased responses in a variety of populations. Moreover, using purified hemagglutinin (HA) vaccines in the form of rDNA-expressed HA protein in a baculovirus expression system has increased immune responses without an increase in reactogenicity. Researchers hypothesize that an increased dosage and 2 doses of a purified influenza vaccine will increase serum hemagglutination inhibition (HAI) and neutralizing antibody responses significantly over those following 2 doses of conventional vaccine in BMT patients. The primary objective of this study is to determine if 2 doses of a baculovirus-expressed recombinant trivalent influenza vaccine containing approximately 135 mcg per HA results in a significantly higher proportion of subjects achieving a Day 28 and Day 56 post vaccination increase in serum HAI and neutralizing antibody titer than seen after immunization with standard dose licensed trivalent inactivated influenza vaccine in immunosuppressed allogeneic HSCT (hematopoietic stem cell transplantation) recipients. The secondary objective is determination of the safety and tolerability of a two-dose regimen of recombinant, baculovirus-expressed HA containing approximately 135 mcg per HA administered by intramuscular injection to patients following allogeneic HSCT, and comparison of the geometric mean titers (GMT) of serum HAI and neutralizing antibody against all 3 virus strains contained in the vaccine. The study will enroll 100 adult (greater than or equal to 18 years of age) allogeneic HSCT recipients between 6 and 12 months following bone marrow transplantation, with no or stable chronic graft-versus-host disease, who are evaluated at the outpatient BMT clinic at M.D. Anderson Cancer Center. Subjects will be randomized to receive either licensed trivalent inactivated influenza vaccine (TIV) or baculovirus-expressed recombinant trivalent hemagglutinin vaccine (rHA0). All injections will be administered into the deltoid muscle. Subjects will be randomized (50 per group) to receive a vaccination on Day 0 and a second dose 4 weeks later. Subjects will be observed in the clinic for at least 20 minutes after inoculation, and subjects will maintain a memory aid to record oral temperature and solicited systemic and local adverse events (AE)s for 8 days (Day 0 through Day 7) after each immunization. Subjects will be seen on Day 2 and Day 30 (1-5 days after each vaccination) for an arm check, vital signs, assessment of possible AEs, concomitant medication assessment, and a targeted physical examination if indicated. Subjects will be contacted by phone on Day 8 and Day 36 (7-10 days after each vaccination) to review the memory aid and to assess for possible AEs or serious (S) AEs. Subjects will return to the clinic on Day 28 for AE and concomitant medication assessment, a targeted physical examination if indicated, and a review of the memory aid prior to receiving the second dose of vaccine. Serum for vaccine immunogenicity evaluations will be collected prior to vaccination at Days 0 and 28, and 56 days after the first vaccine dose. Participants will be involved in study related procedures for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, between 6 and 12 months after undergoing their last allogeneic donor hematopoietic stem cell transplantation with no or stable chronic graft versus host disease (score 0-1).
* Underlying cancer is stable or in complete remission within 3 months prior to enrollment as determined by the treating oncologist in written documentation stating such fact.
* Ambulatory; community dwelling. Subjects will be considered ambulatory if they are not institutionalized, bedridden or homebound.
* Able to return to the clinical site for reactogenicity examinations for at least 7 days after each injection.
* Patients with stable chronic viral infection [(other than Hepatitis B or C and human immunodeficiency virus (HIV)]; any bacterial, mycobacterial or invasive fungal infections that are on maintenance antimicrobial therapy are eligible. Antimicrobial therapy includes: any antiviral, antibacterial or antifungal therapy use under the standard guidelines for treatment or maintenance treatment of viral, bacterial or invasive fungal infections.
* Women of childbearing potential (not surgically sterile or postmenopausal for greater than or equal to 1 year) who are at risk of becoming pregnant must agree to practice adequate contraception (i.e., barrier method, abstinence, or licensed hormonal methods as recommended by her primary care provider) from at least 30 days prior to enrollment and for at least 3 months after receipt of dose 2.
* Able to understand and comply with planned study procedures.
* Provides informed consent prior to initiation of any study procedures and is available for all study visits.

Exclusion Criteria:

* Has moderate or severe chronic graft versus host disease (score 2-3) or uncontrolled chronic graft-versus-host disease (GvHD).
* Has required high-dose corticosteroids: >16 mg prednisone or equivalent daily dose (high-dose methylprednisolone, high-dose dexamethasone), or receiving immunosuppressive agents such as tacrolimus, antithymocyte globulins, cyclosporine, or methotrexate in past 4 weeks.
* Has long-term use (greater than 4 weeks) of moderate to high-dose inhaled steroids (e.g., more than the equivalent of 264 mcg fluticasone; 600 mcg budesonide; 240 mcg beclomethasone; 1000 mcg flunisolide, 750 mcg triamcinolone or 200 mcg mometasone, as a daily dose) within 1 month prior to enrollment.
* Has received chemotherapy within the past 3 months for a refractory or relapsed cancer.
* Was given rituximab or ibritumomab tiuxetan in the past 6 months.
* Splenectomized individuals.
* Has a known allergy to eggs or other components of the vaccine (i.e., thimerosal) or a severe reaction to influenza vaccine in the past.
* Has an acute or chronic condition or an acute change in a chronic condition that (in the opinion of the investigator) would render vaccination unsafe or would interfere with the evaluation of responses including but not limited to the following: acute febrile illness, known chronic liver disease [history of increased alanine transaminase (ALT) and aspartate aminotransferase (AST) levels in the past 4 weeks]; significant renal disease on dialysis; oxygen-dependent chronic lung disease, New York Heart Association Functional Class III or IV; unstable or progressive neurologic disorder; or uncontrolled diabetes mellitus. Medically unstable patients with systolic blood pressure < 90 mmHg, pulse > 100 beats per minutes, or respiratory rate of > 24 per minutes will not be included in this study.
* Has received immunoglobulin within 3 months or monoclonal antibodies within 4 weeks prior to enrollment into the study.
* Has a history of Guillian-Barré Syndrome, vasovagal syncope, clinically symptomatic pericardial effusion or cardiac tamponade, or Bell's palsy.
* Has an acute illness including an oral temperature greater than or equal to 100.0 degrees Fahrenheit, within one week prior to vaccination.
* Has a known history of human immunodeficiency virus (HIV) or Hepatitis B or Hepatitis C. Screening for HIV will not be performed for this study.
* Has a positive urine pregnancy test prior to vaccination (if female of childbearing potential), is breast-feeding, or has the intention to become pregnant within 3 months of receipt of their second dose of vaccine.
* Has received the current licensed trivalent influenza vaccine within the past 4 weeks.
* Has received an investigational agent (drug, vaccine, biologic agent or a device) within 4 weeks before vaccination, or expects to receive an experimental agent prior to completing study visit 5.
* Has a diagnosis of schizophrenia, bipolar disease or other major psychiatric diagnosis.
* Has been hospitalized for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Is receiving psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate). Subjects who are receiving a single antidepressant drug and stable for at least 3 months prior to enrollment, without de-compensating symptoms will be allowed to be enrolled in the study.
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Has any condition that the investigator believes may interfere with successful completion of the study.
* Has a history of alcohol or drug abuse in the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Frequency of four-fold or greater serum hemagglutination inhibition (HAI) and/or neutralization antibody rises in the 2 groups to the 3 hemagglutinin (HA) types (H1, H3, and B) contained within the vaccine. | At Days 28 and 56 after the first vaccine dose.

SECONDARY OUTCOMES:
The frequencies and severity of solicited local and systemic adverse events in each vaccine dosage group. | Day 0 through Day 7 following all vaccinations.
The geometric mean titer (GMT) of serum HAI and serum neutralizing antibody against the influenza A/H3N2, H1N1, and B virus. | 1 month after each vaccination.
The proportion of subjects in each vaccine dose group that achieves a HAI titer of at least 1:32. | 28 days after the first and second dose of vaccine.
Adverse events (AE) or serious adverse events (SAE) information (solicited in-clinic and via memory aids and periodic targeted physical assessment). | Duration of study.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas - MD Anderson Cancer Center - Infectious Diseases, Houston, Texas, United States